CLINICAL TRIAL: NCT01810861
Title: SEROTYPE DISTRIBUTION AND ANTIBIOTIC SUSCEPTIBILITY OF STREPTOCOCCUS PNEUMONIAE CAUSING INVASIVE DISEASES IN CHILDREN AND ADULTS: A LABORATORY- BASED MULTICENTER RETROSPECTIVE STUDY
Brief Title: Serotype Distribution of Streptococcus Pneumoniae That Causes Invasive Diseases at Children and Adults in Turkey
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1851148
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2020-12

CONDITIONS: Pneumococcal Diseases
Keywords: serotype distribution; streptococcus pneumoniae; pneumonia
MeSH Terms: conditions — Pneumococcal Infections; Pneumonia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood, CSF and/or other sterile body areas (catheter, pleural fluid, parasynthesis fluid, pericardial fluid, synovial fluid, BAL)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Serotype distribution (this is a non-interventional study): Serotype distribution both in pediatrics and adults (this is a non interventional study)
  Interventions: Other: There is no intervention in this study

INTERVENTIONS:
Other: There is no intervention in this study — This is a non-interventional study.

SUMMARY:
The aim of this study is to specify the serotype distribution of Streptococcus pneumoniae that causes invasive diseases at children and adults in Turkey.

DETAILED DESCRIPTION:
Non-interventional observational study Descriptive analysis will be conducted.

ELIGIBILITY:
Inclusion Criteria:

Serotype distribution and antibiotic sensitivity of pneumococcal isolates that causes invasive pneumococcal diseases which are obtained from the blood, CSF, and/or all other sterile body areas (catheter, pleural fluid, parasynthesis fluid, pericardial fluid, synovial fluid, BAL) of the adults of 18 years of age or older with children that are younger than 18 years old at these centers and laboratories will be defined.

Exclusion Criteria:

Isolation of any other microorganism than pneumococcus at the same sample.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pneumococcal isolates that are obtained from the blood, CSF and/or other sterile body areas (catheter, pleural fluid, parasynthesis fluid, pericardial fluid, synovial fluid, BAL) with the aim of routine laboratory diagnosis from the pediatric patients that are younger than 18 years old (≤18), who are accepted to the pediatric clinic with the diagnosis of meningitides, bacteremia - sepsis or pneumonia, will be included in the trial.
  S.pneumoniae isolates that meet the inclusion criteria and that are obtained from the invasive clinical samples of the adult patients that are over 18 years old (>18) and applied to the hospital are included in the trial.
Sampling Method: Non-Probability Sample
Enrollment: 922 (Actual)
Dates: Start 2013-01-04 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Identification of S. pneumoniae serotype distribution | 4 years

SECONDARY OUTCOMES:
Identification of antibiotic susceptibility of the isolates | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (32):
- Turkey (Türkiye) (32):
  - Dokuz Eylul University Medical Faculty, Department of Chest Diseases, Balçova, İzmir
  - Ankara Yüksek İhtisas Eğitim ve Araştırma Hastanesi Kardiyoloji Kliniği, Ankara / Altındağ, Turkey
  - Gaziantep Universitesi Tip Fakultesi Mikrobiyoloji, Gaziantep, Turkiye
  - Istanbul Universitesi Istanbul Tip Fakultesi Mikrobiyoloji ve Klinik Mikrobiyoloji Anabilim Dali, Istanbul, Turkiye
  - Cukurova Universitesi Tip Fakultesi Tibbi Mikrobiyoloji Anabilim Dali, Adana
  - Hacettepe Universitesi Tip Fakultesi Cocuk Enfeksiyon Hastaliklari Bilim Dali, Ankara
  - Ankara Meslek Hastalıkları Hastanesi, Ankara
  - Sami Ulus Kadin Dogum Cocuk Sagligi ve Hastaliklari Egitim Arastirma Hastanesi, Ankara
  - Antalya Egitim ve Arastirma Hastanesi Tibbi Mikrobiyoloji, Antalya
  - Akdeniz University Medical Faculty Microbiology Department, Antalya
  - Akdeniz University Medical Faculty, Microbiology, Antalya
  - Samsun Ondokuz Mayis Universitesi Tibbi Mikrobiyoloji ABD, Atakum Samsun
  - Uludag Universitesi Tip Fakultesi Mikrobiyoloji ve Enfeksiyon Hastaliklari Anabilim Dali, Bursa
  - Diyarbakir Dicle Universitesi Tibbi Mikrobiyoloji ABD, Diyarbakır
  - Dicle Universitesi Tip Fakultesi Tibbi Mikrobiyoloji Anabilim Dali, Diyarbakır
  - Firat Universitesi Tip Fakultesi Mikrobiyoloji ve Klinik Mikrobiyoloji Anabilim Dali, Elâzığ
  - Osmangazi University Medical Faculty, Microbiology, Eskişehir
  - Marmara Universitesi Tip Fakultesi, Istanbul
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi Cocuk Sagligi ve Hastaliklari Ana Bilim Dali, Istanbul
  - Ege University Medical Faculty, Microbiology, Izmir
  - İzmir Tepecik Rearch and Training Hospital, Izmir
  - Istanbul Okmeydani Egitim ve Arastirma Hastanesi Kagithane Semt Poliklinii, Kagithane Istanbul
  - Kahramanmaras Sutcu Imam Universitesi Tip Fakultesi Tibbi Mikrobiyoloji Anabilim Dali, Kahramanmaraş
  - Erciyes University Medical Faculty, Kayseri
  - Kayseri Training and Research Hospital, Kayseri
  - Izmir Dr. Behcet Uz Cocuk Hastaliklari ve Cerrahisi Egitim ve Arastirma Hastanesi, Konak Izmir
  - Necmettin Erbakan University Meram Faculty of Medicine Deparment of Pediatrics, Konya
  - Mersin University Medical Faculty, Microbiology, Mersin
  - Hacettepe University Medical Faculty Hospital, Samanpazari, Ankara
  - Selcuk Universitesi Tip Fakultesi Dahili Tip Bilimleri Bolumu Cocuk Sagligi ve Hastaliklari A.B.D, Selcuklu /konya
  - Karadeniz Teknik Universitesi Tip Fakultesi Tibbi Mikrobiyoloji Anabilim Dali, Trabzon
  - Van 100.Yl University Medical Faculty, Van

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1851148&StudyName=Serotype%20Distribution%20And%20Antibiotic%20Susceptibility%20Of%20Streptococcus%20Pneumoniae%20Causing%20Invasive%20Diseases%20In%20Children%20And%20Adults%3A%20A%20Laboratory-%20Based%20Multicenter%20Retrospective%20Study